CLINICAL TRIAL: NCT04994535
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Platysma Prominence
Brief Title: A Study To Assess the Safety and Effects of OnabotulinumtoxinA (BOTOX) Intramuscular Injection in Adult Participants With Platysma Prominence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-310; 2021-000240-22 (EudraCT Number)
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Platysma Prominence
Keywords: Platysma Prominence; OnabotulinumtoxinA; BOTOX
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BOTOX (Experimental): BOTOX (OnabotulinumtoxinA) will be injected into the platysma muscle on Day 1
  Interventions: Drug: OnabotulinumtoxinA
- Placebo (Placebo Comparator): Placebo will be injected into the platysma muscle on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Injection
  Other Names: BOTOX
  Arms: BOTOX
Drug: Placebo — Saline injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and effects of onabotulinumtoxinA (BOTOX) for the temporary improvement in the appearance of platysma prominence.

Study doctors will randomize participants into 1 of the 2 groups, called treatment arms. There is a 1 in 2 chance that a participant will be assigned to placebo. Around 400 participants will be enrolled in the study across approximately 35 sites in USA, Belgium, Canada, Germany and the UK.

Participants will receive a single treatment of intramuscular injection of onabotulinumtoxinA (BOTOX) or placebo on Day 1 during this 4 month long study.

Participants will attend regular monthly visits during the study at the study site.

ELIGIBILITY:
Inclusion Criteria:

* Participants must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study specific procedures
* Are willing and able to comply with procedures required in the protocol
* Adult male or female, at least 18 years old at the time of signing the informed consent
* Good health as determined by medical history, physical examination, vital signs, and investigator's judgment

Exclusion Criteria:

* Any medical condition that may put the participant at increased medical risk with exposure to BOTOX, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* Participant has an anticipated need for treatment with botulinum toxin of any serotype for any indication during the study (other than study intervention)
* Anticipated need for surgery or overnight hospitalization during the study
* Females who are pregnant or breastfeeding and are considering becoming pregnant or donating eggs during the study
* Known immunization or hypersensitivity to any botulinum toxin serotype
* History of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months
* Lower facial and neck hair, scarring (e.g., acne), or other abnormal variations that may interfere with photography (such that photograph is not acceptable)
* Tattoos, jewelry, or clothing that cannot be removed, and that obscure the target area of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (34):
- United States (20):
  - Total Skin and Beauty Derm Ctr /ID# 249905, Birmingham, Alabama
  - Westside Aesthetics /ID# 231196, Los Angeles, California
  - Skin Care and Laser Physicians of Beverly Hills /ID# 231194, Los Angeles, California
  - Moradi MD /ID# 244719, Vista, California
  - Skin Research Institute LLC /ID# 231195, Coral Gables, Florida
  - Skin and Cancer Associates, LLP /ID# 231189, Miami, Florida
  - DeNova Research /ID# 231191, Chicago, Illinois
  - Oak Dermatology in Naperville /ID# 231193, Naperville, Illinois
  - Etre Cosmetic Dermatology and Laser Center /ID# 231192, New Orleans, Louisiana
  - BOYD Beauty Birmingham /ID# 231190, Birmingham, Michigan
  - Michigan Center for Research Corporation /ID# 249911, Clinton Township, Michigan
  - Skin Specialists, PC /ID# 249903, Omaha, Nebraska
  - The Center for Dermatology Cosmetics & Laser Surgery /ID# 231187, Mount Kisco, New York
  - Luxurgery /ID# 244924, New York, New York
  - Coastal Clinical Research Center of the Carolinas /ID# 231197, Charleston, South Carolina
  - Tennessee Clinical Research Center /ID# 244720, Nashville, Tennessee
  - DermResearch, Inc. Austin, TX /ID# 249904, Austin, Texas
  - Bellaire Dermatology Associates /ID# 249902, Bellaire, Texas
  - Austin Institute for Clinical Research at SBA Dermatology /ID# 232104, Houston, Texas
  - Austin Institute for Clinical Research /ID# 244936, Pflugerville, Texas
- Belgium (3):
  - UZ Brussel /ID# 229125, Jette, Brussels Capital
  - Medical Skincare /ID# 229129, Sint-Truiden, Limburg
  - Duinbergen Clinic /ID# 231282, Knokke-Heist, West-Vlaanderen
- Canada (4):
  - Beacon Dermatology Inc /ID# 231675, Calgary, Alberta
  - Pacific Derm /ID# 231019, Vancouver, British Columbia
  - Sweat Clinics of Canada /ID# 231021, Toronto, Ontario
  - Bertucci MedSpa Inc. /ID# 231020, Woodbridge, Ontario
- Germany (5):
  - Studienzentrum Theatiner46 /ID# 229570, Munich, Bavaria
  - Rosenpark Research /ID# 229568, Darmstadt, Hesse
  - Noahklinik GmbH /ID# 232311, Kassel
  - Hautok and Hautok-cosmetics /ID# 229573, München
  - Privatpraxis fuer Dermatologie und Aesthetik /ID# 230901, München
- United Kingdom (2):
  - Waverley Medical Practice /ID# 229590, Coatbridge
  - MediZen Premier Aesthetic Clinic /ID# 229588, Sutton Coldfield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 426 participants were enrolled and randomized into the study (ITT Population); 209 to BOTOX and 217 to placebo. A total of 208 participants were treated with BOTOX and 216 participants were treated with placebo (Safety Analysis Set). A total of 381 participants were included in the modified ITT (mITT) Population; 186 to BOTOX and 195 to placebo. A participant was considered to have completed the study if he/she had at least completed the treatment visit and the end of study visit.
Pre-assignment Details: The ITT Population included all randomized participants; the mITT Population included all randomized participants with a baseline summary score ≥ 19 on the ANLFQ: Impacts questionnaire. The Safety Analysis Set included all participants who were treated with at least 1 dose of study drug.
Groups:
- Placebo: Placebo was injected into the platysma muscle on Day 1
- BOTOX: BOTOX (OnabotulinumtoxinA) was injected into the platysma muscle on Day 1
Period: Overall Study
Arm/Group | Placebo | BOTOX
Started (ITT Population) | 217 | 209
Completed | 199 | 194
Not Completed | 18 | 15
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analyses were performed on the ITT population, consisting of all randomized participants.
Groups:
- BOTOX (onabotulinumtoxinA): BOTOX (onabotulinumtoxinA) was injected into the platysma muscle on Day 1
- Total: Total of all reporting groups
Arm/Group | Placebo | BOTOX (onabotulinumtoxinA) | Total
Number analyzed (Participants) | 217 | 209 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (10.18) | 48.0 (9.57) | 47.5 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 198 | 404
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 30 | 65
  Not Hispanic or Latino | 182 | 179 | 361
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 11 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 202 | 191 | 393
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Time Frame: Enrollment to Day 120
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 216 | 208
Participants | 43 | 34

2. Primary Outcome: Composite Achievement of Grade 1 or 2 (Minimal or Mild) and at Least a 2-Grade Improvement From Baseline Based on Both Investigator's Assessment Using C-APPS and Participant's Self-Assessment Using P-APPS, at Maximum Contraction at Day 14
Description: The Clinician Allergan Platysma Prominence Scale (C-APPS) evaluates platysma prominence severity and is a static measurement encompassing the investigator's visual examination of the platysma muscle at maximum contraction, ranging from 1 - Minimal to 5- Extreme.
  The Participant Allergan Platysma Prominence Scale (P-APPS) evaluates platysma prominence severity and is a single-item measure that is accompanied by a 5-grade photonumeric scale for participants to self-assess the severity of their platysma prominence at maximum contraction, ranging from 1 - Minimal to 5 - Extreme.
Time Frame: Day 14
Population: The intent-to-treat (ITT) population consisted of all randomized participants. Responder rate and its 95% confidence interval (CI) were estimated after using multiple imputation for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants | 0.5 [NA to NA] — NA = Value not estimable due to insufficient number of participants with estimated events after using multiple imputation for missing data. | 31.4 [25.0 to 37.8]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 30.9, 95% CI 2-sided [24.5 to 37.4]

3. Primary Outcome: Achievement of at Least a 2-grade Improvement From Baseline Based on the Investigator's Assessment Using C-APPS at Maximum Contraction at Day 14
Description: The C-APPS evaluates platysma prominence severity and is a static measurement encompassing the investigator's visual examination of the platysma muscle at maximum contraction, ranging from 1 - Minimal to 5- Extreme.
Time Frame: Day 14
Population: The modified intent-to-treat (mITT) population consisted of all randomized participants with a baseline summary score of ≥ 19 for the ANLFQ: Impacts questionnaire. Responder rate and its 95% confidence interval (CI) were estimated after using multiple imputation for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
percentage of participants | 2.2 [0 to 4.3] | 41.0 [33.8 to 48.3]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 38.9, 95% CI 2-sided [31.3 to 46.4]

4. Primary Outcome: Achievement of at Least a 2-grade Improvement From Baseline Based on the Participant's Self-Assessment Using P-APPS at Maximum Contraction at Day 14
Description: The P-APPS evaluates platysma prominence severity and is a single-item measure that is accompanied by a 5-grade photonumeric scale for participants to self-assess the severity of their platysma prominence at maximum contraction, ranging from 1 - Minimal to 5 - Extreme.
Time Frame: Day 14
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
percentage of participants | 3.9 [1.1 to 6.7] | 40.8 [33.5 to 48.1]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 36.9, 95% CI 2-sided [29.1 to 44.7]

5. Secondary Outcome: Percentage of Participants Who Achieved Grade 1 or 2 (Minimal or Mild) According to Investigator's Assessment Using C-APPS at Maximum Contraction at Days 14, 30, 60, 90, and 120
Description: as for outcome 3
Time Frame: Day 14, 30, 60, 90, and 120
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants
  Day 14 | 3.0 [0.6 to 5.3] | 48.3 [41.3 to 55.3]
  Day 30 | 3.3 [0.9 to 5.8] | 43.8 [36.9 to 50.7]
  Day 60 | 4.5 [1.6 to 7.3] | 24.8 [18.8 to 30.8]
  Day 90 | 2.0 [0.1 to 3.9] | 15.2 [10.2 to 20.1]
  Day 120 | 2.5 [0.4 to 4.7] | 14.0 [9.2 to 18.8]

6. Secondary Outcome: Percentage of Participants Who Achieved Grade 1 or 2 (Minimal or Mild) According to Participant's Self-Assessment Using P-APPS at Maximum Contraction at Days 14, 30, 60, 90, and 120
Description: as for outcome 4
Time Frame: Day 14, 30, 60, 90, and 120
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants
  Day 14 | 5.1 [2.1 to 8.2] | 47.1 [40.2 to 54.1]
  Day 30 | 5.6 [2.4 to 8.8] | 41.0 [34.2 to 47.8]
  Day 60 | 7.1 [3.5 to 10.6] | 28.8 [22.4 to 35.2]
  Day 90 | 3.6 [1.0 to 6.2] | 20.6 [14.9 to 26.3]
  Day 120 | 3.8 [1.2 to 6.3] | 16.7 [11.5 to 21.9]

7. Secondary Outcome: Percentage of Participants With Responses of "Satisfied" or "Very Satisfied" on the Appearance of Neck and Lower Face Questionnaire (ANLFQ): Satisfaction (Follow-up) Item 5 (Effect of Treatment) at Day 14
Description: The ANLFQ: Satisfaction scale assesses how satisfied the participants are with the treatment they received for the appearance of their neck and lower face. Item 5 is a verbal descriptor scale ranging from 1 (Very satisfied) to 5 (Very dissatisfied).
Time Frame: Day 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percent of participants | 12.0 [7.4 to 16.5] | 62.1 [55.4 to 68.9]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 50.2, 95% CI 2-sided [42.0 to 58.3]

8. Secondary Outcome: Percentage of Participants With Responses of 'Not at All Bothered' or 'A Little Bothered' on the Bother Assessment Scale - Platysma Prominence (BAS-PP) Scale Item 2 (Jawline) at Day 14
Description: The BAS-PP Scale is a 2-item measure that asks participants to rate how bothered they are by the appearance of their vertical neck bands (Item 1) and jawline (Item 2) where items are rated from 1 (Not at all bothered) to 5 (Extremely bothered).
Time Frame: Day 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants | 23.1 [17.3 to 28.9] | 50.2 [43.3 to 57.1]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 27.1, 95% CI 2-sided [18.1 to 36.1]

9. Secondary Outcome: Percentage of Participants With Responses of 'Not at All Bothered' or 'A Little Bothered' on the BAS-PP Scale Item 1 (Vertical Neck Bands) at Day 14
Description: as for outcome 8
Time Frame: Day 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants | 14.4 [9.5 to 19.2] | 50.2 [43.3 to 57.1]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 35.8, 95% CI 2-sided [27.4 to 44.2]

10. Secondary Outcome: Change From Baseline on the Appearance of Neck and Lower Face Questionnaire (ANLFQ): Impacts Summary Score at Day 14
Description: The ANLFQ: Impacts scale assesses the psychosocial impact due to the appearance of the neck and lower face. All items are rated on a 5-point Verbal Descriptor Scale ranging from 1 (Never) to 5 (All of the time), with higher summary scores (range: 7-35) indicating greater negative psychosocial impact from the appearance of the neck and lower face. For change from baseline in the ANLFQ: Impacts summary score, positive values indicate worsening and negative values indicate improvement in the psychosocial impact.
Time Frame: Day 14
Population: The intent-to-treat (ITT) population consisted of all randomized participants. Least squares mean, its standard error (SE), and its 95% confidence interval (CI) were estimated after using multiple imputation for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
score on a scale | -2.7 (0.45) | -7.1 (0.46)
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < .0001, ANCOVA — P-value derived from ANCOVA model stratified by investigator site and baseline C-APPS with baseline value as a factor; Difference (SE) = -4.4, 95% CI 2-sided [-5.4 to -3.4], Standard Error of Mean 0.51

11. Secondary Outcome: Percentage of Participants Who Achieved at Least 1-Grade Improvement From Baseline Based on Investigator's Assessment Using C-APPS at Maximum Contraction at Days 14, 30, 60, 90, and 120
Description: as for outcome 3
Time Frame: Day 14, 30, 60, 90, and 120
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants
  Day 14 | 20.1 [14.5 to 25.7] | 76.9 [71.0 to 82.7]
  Day 30 | 18.7 [13.2 to 24.3] | 72.6 [66.4 to 78.8]
  Day 60 | 19.5 [13.9 to 25.1] | 54.9 [47.7 to 62.0]
  Day 90 | 17.3 [12.0 to 22.7] | 44.0 [37.0 to 50.9]
  Day 120 | 14.9 [10.0 to 19.9] | 33.9 [27.4 to 40.5]

12. Secondary Outcome: Percentage of Participants Who Achieved at Least 1-Grade Improvement From Baseline Based on Participant's Assessment Using P-APPS at Maximum Contraction at Days 14, 30, 60, 90, and 120
Description: as for outcome 4
Time Frame: Day 14, 30, 60, 90, and 120
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 217 | 209
percentage of participants
  Day 14 | 21.0 [15.3 to 26.6] | 79.3 [73.6 to 84.9]
  Day 30 | 22.8 [17.0 to 28.6] | 73.9 [67.8 to 80.0]
  Day 60 | 20.9 [15.3 to 26.5] | 65.2 [58.6 to 71.9]
  Day 90 | 18.6 [12.9 to 24.2] | 53.7 [46.6 to 60.7]
  Day 120 | 18.8 [13.2 to 24.3] | 42.9 [36.0 to 49.7]

13. Secondary Outcome: Percentage of Participants Who Achieved a Rating of Minimal or Mild According to Participant's Assessment Using P-APPS at Maximum Contraction at Days 14
Description: as for outcome 4
Time Frame: Day 14
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
percentage of participants | 5.2 [1.9 to 8.4] | 48.1 [40.7 to 55.5]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 42.9, 95% CI 2-sided [34.8 to 51.0]

14. Secondary Outcome: Percentage of Participants With Responses of "Satisfied" or "Very Satisfied" on the ANLFQ: Satisfaction (Follow-up) Item 5 (Effect of Treatment) at Day 14
Description: as for outcome 7
Time Frame: Day 14
Population: The modified intent-to-treat (mITT) population consisted of all randomized participants with a baseline summary score of ≥ 19 for the ANLFQ: Impacts questionnaire. Responder rate and its 95% confidence interval (CI) are estimated after using multiple imputation for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
percentage of participants | 11.8 [7.0 to 16.6] | 61.2 [54.0 to 68.4]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 49.4, 95% CI 2-sided [40.8 to 58.1]

15. Secondary Outcome: Percentage of Participants With Responses of 'Not at All Bothered' or 'A Little Bothered' on the BAS-PP Scale Item 2 (Jawline) at Day 14
Description: as for outcome 8
Time Frame: Day 14
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
percentage of participants | 20.6 [14.7 to 26.4] | 49.4 [42.1 to 56.7]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 28.8, 95% CI 2-sided [19.4 to 38.2]

16. Secondary Outcome: Percentage of Participants With Responses of 'Not at All Bothered' or 'A Little Bothered' on the BAS-PP Scale Item 1 (Vertical Neck Bands) at Day 14
Description: as for outcome 8
Time Frame: Day 14
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
percentage of participants | 11.9 [7.2 to 16.6] | 47.8 [40.5 to 55.1]
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) model stratified by investigator site and baseline C-APPS; Difference (%) = 35.9, 95% CI 2-sided [27.2 to 44.6]

17. Secondary Outcome: Change From Baseline on the Appearance of Neck and Lower Face Questionnaire (ANLFQ): Impacts Summary Score at Day 14
Description: as for outcome 10
Time Frame: Day 14
Population: The modified intent-to-treat (mITT) population consisted of all randomized participants with a baseline summary score of ≥ 19 for the ANLFQ: Impacts questionnaire. Least squares mean, its standard error (SE), and its 95% confidence interval (CI) were estimated after using multiple imputation for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
score on a scale | -3.0 (0.50) | -7.7 (0.51)
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Test type: Superiority; p < 0.0001, ANCOVA — P-value derived from ANCOVA model stratified by investigator site and baseline C-APPS with baseline value as a factor; Difference (SE) = -4.7, 95% CI 2-sided [-5.8 to -3.7], Standard Error of Mean 0.54

18. Secondary Outcome: Change From Baseline on the ANLFQ: Impacts Summary Score at Days 30, 60, and 90
Description: The ANLFQ: Impacts scale assesses the psychosocial impact of the appearance of the neck and lower face. All items are rated on a 5-point Verbal Descriptor Scale ranging from 1 (Never) to 5 (All of the time), with higher scores indicating greater negative impact from the appearance of the neck and lower face.
Time Frame: Days 30, 60, and 90
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BOTOX
Number analyzed (Participants) | 195 | 186
score on a scale
  Day 30 | -3.9 (0.54) | -8.8 (0.55)
  Day 60 | -3.5 (0.56) | -8.2 (0.56)
  Day 90 | -3.5 (0.50) | -7.4 (0.50)
Statistical Analysis 1: Comparison: Placebo vs BOTOX; Day 30; Test type: Superiority; p < 0.0001, ANCOVA — P-value derived from ANCOVA model stratified by investigator site and baseline C-APPS with baseline value as a factor; Difference (SE) = -4.9, 95% CI 2-sided [-6.0 to -3.7], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Placebo vs BOTOX; Day 60; Test type: Superiority; p < 0.0001, ANCOVA — P-value derived from ANCOVA model stratified by investigator site and baseline C-APPS with baseline value as a factor; Difference (SE) = -4.7, 95% CI 2-sided [-5.9 to -3.6], Standard Error of Mean 0.59
Statistical Analysis 3: Comparison: Placebo vs BOTOX; Day 90; Test type: Superiority; p < 0.0001, ANCOVA — P-value derived from ANCOVA model stratified by investigator site and baseline C-APPS with baseline value as a factor; Difference (SE) = -3.9, 95% CI 2-sided [-4.9 to -2.8], Standard Error of Mean 0.54

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from enrollment to end of study. The median time participants were followed was 120 days for both the BOTOX and Placebo treatment groups.
Arm/Group | Placebo | BOTOX
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/208
Serious Adverse Events (participants affected / at risk) | 1/216 | 0/208
Other Adverse Events (participants affected / at risk) | 6/216 | 7/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=216) | BOTOX (N=208)
ADNEXA UTERI CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=216) | BOTOX (N=208)
COVID-19 (Infections and infestations) | 6 (6) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04994535/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT04994535/SAP_001.pdf